CLINICAL TRIAL: NCT04590417
Title: Institute of HIV Research and Innovation (IHRI)
Brief Title: Assessment of Drug-drug Interactions Between Feminizing Hormone Therapy and Emtricitabine/Tenofovir Alafenamide Concomitantly for Pre-exposure Prophylaxis Among Transgender Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: iFACT 3
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Estradiol; Cyproterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 HIV-negative TGW (Other): A single-arm prospective PK study of HIV-negative TGW taking FHT and daily PrEP.
  Interventions: Drug: Estradiol valerate 2 mg, cyproterone acetate 25 mg

INTERVENTIONS:
Drug: Estradiol valerate 2 mg, cyproterone acetate 25 mg — The entire study period will be approximately 1 year, which will include around 2 months of document preparation, 5 months of recruitment, 3 months of follow-up, and 2 months of data analysis.

SUMMARY:
Recent studies have showed that there were significant drug-drug interactions (DDI) from feminizing hormone therapy (FHT) towards emtricitabine/tenofovir disoproxil fumarate (F/TDF)-based pre-exposure prophylaxis (PrEP) among transgender women (TGW). New strategies for PrEP among TGW who use FHT are urgently needed. Because tenofovir alafenamide (TAF) can achieve higher intracellular TFV-DP levels with lower tenofovir plasma concentrations, it is promising that both plasma TFV and intracellular TFV-DP levels might not be significantly affected by FHT. The current study aims to determine the pharmacokinetics DDI between FHT and F/TAF-based PrEP among TGW.

DETAILED DESCRIPTION:
Two full pharmacokinetic (PK) measurements will be performed. Samples collected will include: plasma for estradiol (E2), emtricitabine (FTC), tenofovir (TFV), and tenofovir alafenamide (TAF) measurement; and peripheral blood mononuclear cells (PBMC) for emtricitabine-triphosphate (FTC-TP) and tenofovir-diphosphate (TFV-DP) intracellular quantification.

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Age 18-40 years old
3. Transgender women
4. HIV-negative
5. Body mass index 18.5-24.9 kg/m2
6. Calculated creatinine clearance (CrCl) ≥60 mL/min, as estimated by the Cockcroft-Gault equation
7. Alanine aminotransferase (ALT) ≤2.5 x ULN
8. Signed the informed consent form

Exclusion Criteria:

1. Known history of allergy to hormonal component to be used in the study
2. Male-to-female transgender who underwent orchiectomy
3. Use of pre-exposure prophylaxis or post-exposure prophylaxis in the past 30 days
4. Use of injectable FHT in the past 3 months
5. Evidence of current hepatitis B virus infection (HBV) - i.e. hepatitis B surface antigen (HBsAg) positive
6. Evidence of current hepatitis C virus infection (HCV) - i.e. HCV antibody positive
7. Current use of any of the following:

   * Anticonvulsants: carbamazepine, felbamate, oxcarbazepine, phenytoin, phenobarbital, primidone or topiramate
   * Herbs: gingko biloba, St John's wort or milk thistle
   * Anti-infective agents: azole antifungals, macrolides, griseofulvin, protease inhibitors, rifampicin or rifabutin
8. Participant-reported active rectal infection requiring treatment
9. History of gastrointestinal tract surgery that alter gastrointestinal tract and/or drug absorption
10. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma estradiol levels | Measured at week 3 and week 9 of the study period
Changes in plasma PrEP levels | Week 9 through 12
  1. Plasma TFV
  2. Plasma FTC
  3. Plasma TAF
Changes in intracellular PrEP levels | Week 9 through 12
  1. PBMC TFV-DP levels
  2. PBMC FTC-TP levels

SECONDARY OUTCOMES:
Changes in plasma testosterone levels | Week 3 through 9

CONTACTS AND LOCATIONS:
Overall Officials: Siriporn Nonenoy, RN.MPH., Study Chair — Institute of HIV Research and Innovation (IHRI)
Locations (1):
- Institute of HIV Research and Innovation (IHRI), Bangkok, Pathumwan, Thailand

REFERENCES:
- [Derived] Hiransuthikul A, Thammajaruk N, Kerr S, Janamnuaysook R, Nonenoy S, Hongchookiat P, Trichavaroj R, Tawon Y, Boonruang J, Teeratakulpisarn N, Cressey TR, Anderson PL, Phanuphak N; iFACT3 study team. No significant drug-drug interaction between oral TAF-based PrEP and feminizing hormone therapy among transgender women in Thailand: the iFACT-3 study. J Int AIDS Soc. 2025 May;28(5):e26502. doi: 10.1002/jia2.26502. PMID 40390323